CLINICAL TRIAL: NCT00341549
Title: Family Myopia Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902191; 02-HG-N191
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Myopia
Keywords: Genetics; Mapping; Gene; Myopia; Nearsightedness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Myopia: The subject population will be adult individuals and their children, in good health with the exception of myopia.

SUMMARY:
This study will try to identify the gene or genes responsible for myopia (nearsightedness) and to examine the relationship between myopia and near work. Myopia is the most common eye disorder in the world, affecting one in four Americans. Several studies indicate that myopia is inherited. The condition tends to cluster in families, so that studying families with this condition may facilitate finding the exact cause.

Caucasian Americans and African Americans with myopia who are in general good health may be eligible for this study. People with a family history of myopia through several generations along one parent s side only, and in which more than one sibling has myopia are preferred. People who have severe diseases that involve myopia, such as Stickler s or Marfan syndromes, retinitis pigmentosa or diabetic retinopathy may not participate.

Participants will undergo the following tests and procedures:

* Eye examination, including refraction
* Blood draw for genetic studies and possibly establishment of cell lines (collection of cells grown in the laboratory from an original tissue specimen) for future research
* Myopia Family Study Questionnaire and personal medical information questionnaire to provide information about other medical conditions that may influence the development of myopia; the vision status of their spouse and children, parents and siblings, and spouse s parents and siblings
* Risk Factor Questionnaire (for Jewish Orthodox community only) to assess the amount of near work activity done in childhood

DETAILED DESCRIPTION:
Myopia or nearsightedness, a condition that results in the inability to see distant objects clearly, affects one in four Americans and is the most common eye disorder in the world with an enormous public health and economic impact. Depending on epidemiologic definition, 3-19% of acquired blindness has been ascribed to myopia. Evidence exists that myopia is a complex disorder with a significant genetic component as well as potential environmental influences. Implicating genetic factors, Sorsby et al. found that the trait correlation for monozygotic twins was nearly twice that for dizygotic twins and zero for control pairs. A study, by Chen et al., of Chinese twin pairs found a higher concordance rate of myopia (92.2%) for monozygotic twins with concordant close-work habits, or differences of less than one hour per day spent studying or reading, as compared to monozygotic twins with discordant close-work habits (79.3%). The two studies suggest additive interaction between zygosity and close-work habits.

Since there is a tendency of myopia to cluster in families, studying families with myopia opens the possibility to identify any gene(s) responsible for the pathogenesis of myopia. These genes could provide molecular tools for investigation of inherited myopia and may also provide a starting point for elucidating mechanisms for the influence of near work on the progression of myopia. The goal of this proposal is to identify regions of the human genome that contain the genes responsible for non-syndromic myopia utilizing pedigrees identified by the Myopia Family Study and genotypes generated by Dr. Dwight Stambolian's laboratory at the University of Pennsylvania as well as by the Center for Inherited Disease Research. Pedigree collection is ongoing in several geographic regions including Lakewood, NJ, for the collection of Orthodox Jewish families, Lancaster County, PA for the collection of Amish families, and Philadelphia, for recruitment of families of African American or Chinese American background. Pedigrees of Caucasian descent have also been collected in Philadelphia. All data collection is under the direction of Dr. Stambolian and funded by his grant from the NEI; no NHGRI funds are being used for data collection, and NHGRI investigators do not have any contact with study subjects. Because this disorder is complex and has a high likelihood of being caused by multiple loci, multiple parametric and non-parametric methods of analysis will be employed. Heterogeneity will be taken into account during these analyses, as will environmental covariates, such as the effect of near work, when possible.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subject population will be adult individuals and their children, in good health with the exception of myopia.

Subjects will be chosen based upon vision history of their extended family.

Preferred subjects will be those who have a family in which myopia passes through several generations along one parent s side only, in which more than one sibling is affected with myopia, but in which no more than one parent is affected.

Specific eligibility requirements for the index case include:

1. Cycloplegic refraction of 1.00 spherical equivalent (as long as there was 1.00D or higher in each meridian if astigmatism is present) or worse in both eyes in those under age 50 to be considered myopic;
2. Manifest refraction of 1.00 spherical equivalent (as long as there was 1.00D or higher in each meridian if astigmatism is present) or worse in both eyes in those over age 50 to be considered myopic;
3. No history of systemic or ocular disease which might predispose to myopia including premature birth;
4. The index case should have a familial history of myopia in either their parents or children or other close relatives (suggesting a genetic influence);
5. In the event that the parents of the index case have myopia, it is preferred that only one parent be affected with myopia.

Some of these bilineal families may be collected if necessary to achieve the desired sample size, but unilateral families are preferred.

EXCLUSION CRITERIA:

Excluded from the University of Pennsylvania study are those who have severe diseases that involve myopia, such as Stickler s or Marfan syndromes, ocular disease such as Retinitis Pigmentosa, and those with diseases that may secondarily cause myopia such as diabetes or retinopathy of prematurity. Records of eye examinations obtained prior to the onset of systemic or ocular disease will be accepted.

Individuals who complete the Risk Factor Questionnaire and who state that they were born more than a month prematurely will not be included in the study.

Individuals who are myopic in one eye and unaffected in the other (ulnilateral myopes) will not be included in the study.

Individuals who do not sign the Consent Form will be excluded, and families for whom all necessary members do not sign the Consent Form will be excluded.

No fetuses, pregnant women, prisoners or other institutionalized individuals will be enrolled.

Generally, myopia itself is not associated with mental impairment, although careful consideration will be given to determining the cognitive understanding of any such potentially impaired person appropriate for enrollment in order to assure that protection of human rights is optimized.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population will be adult individuals and their children, in good health with the exception of myopia.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 7477 (Actual)
Dates: Start 2002-04-29 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Myopia Genes | Ongoing
  The overall objective for this project is to query the entire human genome to identify the genes responsible for myopia and for variation in ocular refraction.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bailey-Wilson, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young TL, Ronan SM, Drahozal LA, Wildenberg SC, Alvear AB, Oetting WS, Atwood LD, Wilkin DJ, King RA. Evidence that a locus for familial high myopia maps to chromosome 18p. Am J Hum Genet. 1998 Jul;63(1):109-19. doi: 10.1086/301907. PMID 9634508
- [Background] Young TL, Ronan SM, Alvear AB, Wildenberg SC, Oetting WS, Atwood LD, Wilkin DJ, King RA. A second locus for familial high myopia maps to chromosome 12q. Am J Hum Genet. 1998 Nov;63(5):1419-24. doi: 10.1086/302111. PMID 9792869
- [Background] Sperduto RD, Seigel D, Roberts J, Rowland M. Prevalence of myopia in the United States. Arch Ophthalmol. 1983 Mar;101(3):405-7. doi: 10.1001/archopht.1983.01040010405011. PMID 6830491